CLINICAL TRIAL: NCT03398512
Title: A Study of Conversion Therapy Using Hyperthermic Intraperitoneal Chemoperfusion (HIPEC) and Systemic Oxaliplatin/Capecitabine Chemotherapy in Unresectable Peritoneal Metastases From Colorectal Cancer
Brief Title: HIPEC and Systemic Chemotherapy in Unresectable Peritoneal Metastases From Colorectal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrolled patients received the second surgery.
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Bin Xiong, MD, Zhongnan Hospital, Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WuhanU_Peritoneal M_colon
Record Dates: First submitted 2018-01-04; First posted 2018-01-12 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Peritoneal Metastases From Colorectal Cancer
MeSH Terms: interventions — Laparotomy; Hyperthermic Intraperitoneal Chemotherapy; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): HIPEC with Raltitrexed at the time of fist surgery and twice repeat within one week after the surgery, following 3 cycles of 3-week Oxaliplatin/Capecitabine chemotherapy. The second surgery, exploratory laparoscopy or laparotomy, is carried out one week later after the series of systemic chemotherapy.
  Interventions: Procedure: exploratory laparoscopy or laparotomy; Procedure: HIPEC; Drug: Systemic chemotherapy

INTERVENTIONS:
Procedure: exploratory laparoscopy or laparotomy — Exploratory laparoscopy or laparotomy, for PCI score or radical colorectal resection and cytoreductive surgery
Procedure: HIPEC — Normal saline 3000ml-4000ml, Raltitrexed 4mg, 43°C, 60min.
Drug: Systemic chemotherapy — Oxaliplatin: 130mg/m2, day 1. Capecitabine: 1500mg, twice daily for two weeks, and then suspend for one week

SUMMARY:
The prognosis of patients with unresectable peritoneal metastases from colorectal cancer is poor. These patients may obtain survival benefit from radical colorectal resection and cytoreductive surgery (CRS). The response rates of previous conversion therapy are low. Hyperthermic intraperitoneal chemoperfusion (HIPEC) and systemic chemotherapy are effective methods of reducing peritoneal cancer index (PCI) levels. The purpose of this study is to investigate the efficacy and safety of HIPEC and systemic chemotherapy in the conversion therapy of peritoneal metastases from colorectal cancer.

DETAILED DESCRIPTION:
To determine the efficacy and safety of HIPEC and systemic chemotherapy in the conversion therapy of peritoneal metastases from colorectal cancer, patients undergo HIPEC with Raltitrexed at the time of fist surgery and twice repeat within one week after the surgery, following 3 cycles of 3-week Oxaliplatin/Capecitabine chemotherapy. The second surgery, exploratory laparoscopy or laparotomy, is carried out one week later after the series of systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological proved diagnosis of colorectal cancer.
* Unresectable peritoneal metastases and primary tumor proved at surgery.
* No evidence of distant metastases.
* Have not received radiotherapy, chemotherapy or immunotherapy.
* ECOG score: 0~2.
* Written informed consent is obtained prior to commencement of trial treatment.

Exclusion Criteria:

* Existence of distant metastasis outside the abdomen.
* Any previous radiotherapy, chemotherapy or immunotherapy.
* Active systemic infections.
* Inadequate cardiac function, renal function, liver function or bone marrow function at the beginning of the trial.
* Female patients who are pregnant or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
radical resection rate | 3 months
  The rate between the number of patients with radically resectable peritoneal metastases and those with unresectable peritoneal metastases

SECONDARY OUTCOMES:
the Peritoneal Cancer Index score | 3 months
  The score range from 0 to 39, higher values represent a worse outcome
overall survival | 3 years
  The overall survival time
complication rate | 3 years
  The rate of adverse complication

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan University, Wuhan, Hubei, China